CLINICAL TRIAL: NCT02256553
Title: A Phase IV, Open-label, Safety and Tolerability Trial of MK-3641 and MK-7243 Coadministered in Subjects At Least 18 Years of Age With Ragweed and Grass Pollen Induced Allergic Rhinitis With or Without Conjunctivitis
Brief Title: Safety Study of MK-3641 and MK-7243 Co-administered in Adult Participants With Ragweed and Grass Pollen Induced Allergic Rhinitis (P08607, MK-3641-006)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: ALK-Abelló A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P08607
Record Dates: First submitted 2014-10-01; First posted 2014-10-03 (Estimated); Results first posted 2016-01-18 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-01

CONDITIONS: Rhinitis, Allergic, Seasonal
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MK-3641+ MK-7243 (Experimental): Participants receive one MK-7243 tablet, SL QD in the evening for 14 days during Period I; one MK-3641 tablet, SL QD in the morning and one MK-7243 tablet, SL QD in the evening for 14 days during Period II; and one MK-3641 tablet, SL QD, and one MK-7243 tablet, SL QD, within 5 minutes of each other for 14 days during Period III.
  Interventions: Biological: MK-3641 12 Amb a 1-U (short ragweed extract); Biological: MK-7243 2800 BAU (Timothy grass extract); Drug: Rescue Medication

INTERVENTIONS:
Biological: MK-3641 12 Amb a 1-U (short ragweed extract) — 12 units of Ambrosia artemisiifolia major allergen number 1 (Amb a 1-U) extract sublingual tablets
  Other Names: SCH 039641; RAGWITEK®
Biological: MK-7243 2800 BAU (Timothy grass extract) — 2800 bioequivalent allergen units (BAU) of Phleum pratense extract sublingual tablets
  Other Names: SCH 697243; GRASTEK®
Drug: Rescue Medication — Self-injectable epinephrine, to be administered for an anaphylactic reaction, including symptoms/signs of upper airway obstruction.

SUMMARY:
The purpose of this study is to assess the safety and tolerability of MK-3641 (short ragweed [Ambrosia artemisiifolia] extract, SCH 039641, RAGWITEK®) sublingual tablets and MK-7243 (Timothy grass [Phleum pratense] extract, SCH 697243, GRASTEK®) sublingual tablets co-administered in participants 18 through 65 years of age with both ragweed- and grass polled-induced allergic rhinitis, with or without conjunctivitis and with or without asthma. The primary endpoint is the percentage of participants who experience at least one event of local swelling after co-administration of MK-3641 and MK-7243 sublingual tablets.

DETAILED DESCRIPTION:
Events of local swelling include pharyngeal edema, laryngeal edema, mouth edema, oropharyngeal swelling, palatal edema, tongue swelling/edema or throat tightness.

ELIGIBILITY:
Inclusion Criteria:

* Clinical history of physician-diagnosed ragweed- and grass pollen-induced rhinitis with or without conjunctivitis of >1 year duration, with or without asthma
* Female participants of childbearing potential must have a negative urine pregnancy test at Screening and Randomization Visits and must agree to remain abstinent or use (or have their partner use) any one of the acceptable methods of birth control within the projected duration of the study. Acceptable methods of birth control are: intrauterine device (IUD), diaphragm with spermicide, contraceptive sponge, condom, vasectomy, hormonal contraception.

Exclusion Criteria:

* Unstable, uncontrolled or severe asthma treated with long-acting beta agonists (LABAs) at the time of Screening
* Received immunosuppressive treatment within 3 months prior to Randomization (except steroids for allergic reactions other than asthma)
* History of anaphylaxis with cardiorespiratory symptoms with prior immunotherapy, unknown cause, or inhalant allergen
* Diagnosis of eosinophilic esophagitis
* History of any severe systemic allergic reaction or any severe local reaction to sublingual allergen immunotherapy
* Female and breastfeeding, pregnant or intending to become pregnant
* Received another form of allergen immunotherapy with the past month
* Previously exposed to MK-3641 (RAGWITEK®) or other sublingual ragweed immunotherapy
* Previously exposed to MK-7243 (GRASTEK®) or other sublingual grass immunotherapy
* Known history of allergy, hypersensitivity, or intolerance to the excipient ingredients of the study drug (except for Ambrosia artemisiifolia and/or Phleum pratense), or self-injectable epinephrine
* Unable to or will not comply with the use of self-injectable epinephrine
* Used an investigational drug within 30 days prior to Screening Visit, or plans to participate in another interventional clinical trial during the duration of this trial
* Family member of the investigational or sponsor staff involved in this trial
* Participating in this same trial at another investigational site.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2014-10; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Maloney J, Berman G, Gagnon R, Bernstein DI, Nelson HS, Kleine-Tebbe J, Kaur A, Li Q, Nolte H. Sequential Treatment Initiation with Timothy Grass and Ragweed Sublingual Immunotherapy Tablets Followed by Simultaneous Treatment Is Well Tolerated. J Allergy Clin Immunol Pract. 2016 Mar-Apr;4(2):301-9.e2. doi: 10.1016/j.jaip.2015.11.004. Epub 2016 Jan 2. PMID 26755098

RESULTS

PARTICIPANT FLOW:
Groups:
- MK-3641+MK-7243: Participants receive one MK-7243 tablet, sublingually (SL) once a day (QD) in the evening for 14 days during Period I; one MK-3641 tablet, SL QD in the morning and one MK-7243 tablet, SL QD in the evening for 14 days during Period II; and one MK-3641 tablet, SL QD, and one MK-7243 tablet, SL QD, within 5 minutes of each other for 14 days during Period III.
Period: Period I
Arm/Group | MK-3641+MK-7243
Started | 102
Completed | 96
Not Completed | 6
Not completed — Adverse Event | 5
Not completed — Protocol Violation | 1
Period: Period II
Arm/Group | MK-3641+MK-7243
Started | 96
Completed | 94
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Subject Moved | 1
Period: Period III
Arm/Group | MK-3641+MK-7243
Started | 94
Completed | 91
Not Completed | 3
Not completed — Adverse Event | 3

BASELINE CHARACTERISTICS:
Groups:
- MK-3641+MK-7243: Participants receive one MK-7243 tablet, SL QD in the evening for 14 days during Period I; one MK-3641 tablet, SL QD in the morning and one MK-7243 tablet, SL QD in the evening for 14 days during Period II; and one MK-3641 tablet, SL QD, and one MK-7243 tablet, SL QD, within 5 minutes of each other for 14 days during Period III.
Arm/Group | MK-3641+MK-7243
Number analyzed (Participants) | 102
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.0 (12.0)
Gender [Count of Participants; unit: Participants]
  Female | 53
  Male | 49

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Experienced at Least One Event of Local Swelling
Description: Events of local swelling included pharyngeal edema, laryngeal edema, mouth edema, oropharyngeal swelling, palatal edema, tongue swelling/edema, or throat tightness. Events that occurred during in-clinic dosing were to be monitored and recorded by clinic staff. A Side Effect Report Card was used in Periods I-III to collect information on adverse events identified by the World Allergy Organization (WAO) as local side effects of sublingual immunotherapy (SLIT) that occurred within the first 60 minutes after study drug intake. During Period I, participants were to complete the report card once a day after MK-7243 was administered. During Period II, participants were to complete the report card twice a day, once after each tablet was administered. During Period III, participants were to complete the report card once a day after both tablets were administered.
Time Frame: During Period I, Period II and Period III (Up to 6 weeks)
Population: All Treated Participants population consisted of all participants who received ≥1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | MK-3641+MK-7243
Number analyzed (Participants) | 102
Percentage of Participants
  Period I | 13.7 [7.7 to 22.0]
  Period II | 21.6 [14.0 to 30.8]
  Period III | 14.7 [8.5 to 23.1]

2. Secondary Outcome: Percentage of Participants Who Experienced at Least One Event of Local Application Site Reaction
Description: Events of local application site reactions included pharyngeal edema, laryngeal edema, mouth edema, oropharyngeal swelling, palatal edema, tongue swelling/edema, throat tightness, lip swelling/edema, ear pruritus, dysphagia, oral discomfort, glossodynia, oral pruritus, hypoaesthesia oral, throat irritation, paraesthesia oral or stomatitis. Events that occurred during in-clinic dosing were to be monitored and recorded by clinic staff. A Side Effect Report Card was used in Periods I-III to collect information on adverse events identified by the WAO as local side effects of SLIT that occurred within the first 60 minutes after study drug intake. During Period I, participants were to complete the report card once a day after MK-7243 was administered. During Period II, participants were to complete the report card twice a day, once after each tablet was administered. During Period III, participants were to complete the report card once a day after both tablets were administered.
Time Frame: During Period I, Period II and Period III (Up to 6 weeks)
Population: All Treated Participants population consisted of all participants who received ≥1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | MK-3641+MK-7243
Number analyzed (Participants) | 102
Percentage of Participants
  Period I | 70.6 [60.7 to 79.2]
  Period II | 68.6 [58.7 to 77.5]
  Period III | 55.9 [45.7 to 65.7]

3. Secondary Outcome: Percentage of Participants Who Discontinued Study Drug Due to an Adverse Event (AE)
Description: An AE was defined as any unfavorable and unintended sign, symptom, or disease temporally associated with the use of study drug, whether or not considered related to the study drug. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition that is temporally associated with the use of the study drug, was also an AE.
Time Frame: During Period I, Period II and Period III (Up to 6 weeks)
Population: All Treated Participants population consisted of all participants who received ≥1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | MK-3641+MK-7243
Number analyzed (Participants) | 102
Percentage of Participants
  Period I | 4.9 [1.6 to 11.1]
  Period II | 1.0 [0.0 to 5.3]
  Period III | 2.9 [0.6 to 8.4]

4. Secondary Outcome: Percentage of Participants Who Experienced at Least One Local Application Site Reaction That Required Symptomatic Treatment
Description: as for outcome 2
Time Frame: During Period I, Period II and Period III (Up to 6 weeks)
Population: All Treated Participants population consisted of all participants who received ≥1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | MK-3641+MK-7243
Number analyzed (Participants) | 102
Percentage of Participants
  Period I | 4.9 [1.6 to 11.1]
  Period II | 3.9 [1.1 to 9.7]
  Period III | 1.0 [0.0 to 5.3]

ADVERSE EVENTS:
Time Frame: Up to 8 weeks
Description: All Treated Participants population consisted of all participants who received ≥1 dose of study drug.
Groups:
- Period I: MK-7243; Period II: MK-3641+MK-7243; Period III: MK-3641+MK-7243: Participants receive one MK-7243 tablet, SL QD in the evening for 14 days during Period I; one MK-3641 tablet, SL QD in the morning and one MK-7243 tablet, SL QD in the evening for 14 days during Period II; and one MK-3641 tablet, SL QD, and one MK-7243 tablet, SL QD, within 5 minutes of each other for 14 days during Period III.
Arm/Group | Period I: MK-7243 | Period II: MK-3641+MK-7243 | Period III: MK-3641+MK-7243
Serious Adverse Events (participants affected / at risk) | 0/102 | 1/96 | 0/94
Other Adverse Events (participants affected / at risk) | 74/102 | 68/96 | 55/94
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Period I: MK-7243 (N=102) | Period II: MK-3641+MK-7243 (N=96) | Period III: MK-3641+MK-7243 (N=94)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Period I: MK-7243 (N=102) | Period II: MK-3641+MK-7243 (N=96) | Period III: MK-3641+MK-7243 (N=94)
Ear pruritus (Ear and labyrinth disorders) | 34 (66) | 33 (68) | 20 (38)
Abdominal pain upper (Gastrointestinal disorders) | 7 (8) | 11 (21) | 6 (10)
Glossodynia (Gastrointestinal disorders) | 8 (9) | 9 (13) | 7 (13)
Lip swelling (Gastrointestinal disorders) | 12 (13) | 14 (19) | 10 (13)
Mouth ulceration (Gastrointestinal disorders) | 7 (7) | 7 (9) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 8 (19) | 0 (0)
Oedema mouth (Gastrointestinal disorders) | 0 (0) | 6 (11) | 9 (15)
Oral pruritus (Gastrointestinal disorders) | 51 (95) | 46 (109) | 33 (54)
Palatal oedema (Gastrointestinal disorders) | 0 (0) | 7 (8) | 0 (0)
Paraesthesia oral (Gastrointestinal disorders) | 6 (7) | 0 (0) | 0 (0)
Swollen tongue (Gastrointestinal disorders) | 0 (0) | 10 (13) | 0 (0)
Tongue ulceration (Gastrointestinal disorders) | 8 (9) | 0 (0) | 0 (0)
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 9 (12) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 0 (0) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 54 (93) | 45 (99) | 29 (46)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this study 45 days prior to submission for publication/presentation.